CLINICAL TRIAL: NCT02154334
Title: An Open-label Study to Assess the Effects of Allergic Rhinitis and Coadministration of Mometasone or Oxymetazoline on the Pharmacokinetics, Safety, and Tolerability of Intranasal Esketamine
Brief Title: Study to Assess the Effects of Allergic Rhinitis and Co-administration of Mometasone or Oxymetazoline on the Pharmacokinetics, Safety, and Tolerability of Intranasal Esketamine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR104359; ESKETINTRD1007 (Other: Janssen Research and Development, LLC); 2014-000534-38 (EudraCT Number)
Record Dates: First submitted 2014-05-30; First posted 2014-06-03 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Allergic Rhinitis
Keywords: Allergic Rhinitis; Healthy; Esketamine; Mometasone; Oxymetazoline; Phase 1
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Esketamine; Mometasone Furoate; Oxymetazoline

ARMS (3):
- Cohort 1 (Experimental): One Intranasal spray of 14 milligram (mg) esketamine solution in each nostril on Day 1 at time 0 and 5 minutes (total esketamine dose will be 56 mg) in Period 1 (Treatment A). Two intranasal sprays of 50 microgram (mcg) mometasone suspension in each nostril for a total dose of 200 mcg on days 1 to 15 and 2 intranasal sprays of 50 mcg mometasone suspension in each nostril for a total dose of 200 mcg at time -1 hour prior to 1 intranasal spray of 14 mg esketamine solution in each nostril at time 0 and 5 minutes, for a total dose of 56 mg on Day 16 in Period 2 (Treatment B).
  Interventions: Drug: Esketamine; Drug: Mometasone
- Cohort 2: Sequence 1 (Experimental): One Intranasal spray of 14 mg esketamine solution in each nostril at time 0 and 5 minutes (total esketamine dose will be 56 mg) in Period 1 (Treatment A) and pretreatment with 2 sprays of oxymetazoline 0.05 percent (%) weight by volume (w/v) solution in each nostril at time -1 hour before administration of 1 Intranasal spray of 14 mg esketamine solution in each nostril at time 0 and 5 minutes, for a total dose of 56 mg in Period 2 (Treatment C).
  Interventions: Drug: Esketamine; Drug: Oxymetazoline
- Cohort 2: Sequence 2 (Experimental): Pretreatment with 2 sprays of oxymetazoline 0.05 percent (%) weight by volume (w/v) solution in each nostril at time -1 hour before administration of 1 Intranasal spray of 14 mg esketamine solution in each nostril at time 0 and 5 minutes, for a total dose of 56 mg in Period 1 (Treatment C) and 1 Intranasal spray of 14 mg esketamine solution in each nostril at time 0 and 5 minutes (total esketamine dose will be 56 mg) in Period 2 (Treatment A).
  Interventions: Drug: Esketamine; Drug: Oxymetazoline

INTERVENTIONS:
Drug: Esketamine — Participants will self-administer one Intranasal spray of 14 mg esketamine solution in each nostril on Day 1 at time 0 and 5 minutes (total esketamine dose will be 56 mg) in Period 1 and Period 2.
Drug: Mometasone — Healthy participants will self-administer 2 intranasal sprays of 50 mcg mometasone suspension in each nostril for a total dose of 200 mcg on days 1 to 15 and 2 intranasal sprays of 50 mcg mometasone suspension in each nostril prior to 1 intranasal spray of esketamine solution 14 mg in each nostril at Time 0 and 5 minutes for a total dose of 56 mg on Day 16 in Period 2.
  Arms: Cohort 1
Drug: Oxymetazoline — Nasal rhinitis participants will self-administer 2 intranasal sprays of Oxymetazoline 0.05% w/v solution in each nostril at time -1 hour before administration of 1 Intranasal spray of 14 mg esketamine solution in each nostril at time 0 and 5 minutes, for a total dose of 56 mg in Period 1or Period 2.
  Arms: Cohort 2: Sequence 1; Cohort 2: Sequence 2

SUMMARY:
The purpose of this study is to evaluate the effects of allergic rhinitis (group of symptoms affecting the nose) and co-administration of mometasone or oxymetazoline on the pharmacokinetics (explores what the body does to the drug), safety, and tolerability of intranasal (administered through the nose) esketamine.

DETAILED DESCRIPTION:
This is a Phase 1, single-center, open -label (all people know the identity of the intervention) study of intranasal esketamine in two cohorts: Cohort 1 will be healthy participants assigned to a fixed treatment sequence and Cohort 2 will be participants with nasal rhinitis randomized to 1 of 2 treatment sequences. For all participants, the study comprises 3 phases: a Screening phase (up to 21 days), an Open Label Treatment phase (includes 2 treatment periods; Period 1 and Period 2) and Follow-up phase (10 +/-2 days after last dose of esketamine).

Total study duration for participants in Cohort 1 is up to 52 days which includes Screening phase, Period 1 (3 days) where participants will self-administer a 56 milligram (mg) intranasal dose of esketamine solution on Day 1 and Period 2 (16 days) where participants will self-administer 200 microgram (mcg) of intranasal mometasone suspension on Day 1 (which will begin immediately following the 30 hour pharmacokinetic sample of Period 1) to Day 15, and then 200 mcg of intranasal mometasone suspension prior to a 56 mg dose of intranasal esketamine solution on Day 16 and the follow-up phase. Total study duration for participants in Cohort 2 is up to 44 days which includes Screening phase, Period 1 and Period 2 each of 3 days with a washout period of 5 to 10 days in-between esketamine dosing, and the follow-up phase. Cohort 2 participants will be randomly assigned to either treatment Sequence 1 or 2, wherein Sequence 1 comprises a 56 mg intranasal dose of esketamine solution alone in period 1 followed by period 2 which comprises a pretreatment with oxymetazoline 0.05 percent (%) weight by volume (w/v) solution 1 hour before administration of a 56 mg intranasal dose of esketamine solution. Sequence 2 comprises of a pretreatment with oxymetazoline 0.05 % w/v solution 1 hour before administration of a 56 mg intranasal dose of esketamine solution in Period 1 followed by period 2 which comprises a 56 mg intranasal dose of esketamine solution alone. Blood samples will be collected for evaluation of pharmacokinetic parameters of intranasal esketamine in healthy participants and participants with allergic rhinitis. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Female participant must be postmenopausal (no spontaneous menses for at least 2 years), surgically sterile, abstinent (abstinence is an acceptable means of birth control only if it is already established as the participant's usual and preferred lifestyle), or, if sexually active, be practicing an effective method of birth control (for example, prescription oral contraceptives, contraceptive injections, intrauterine device, double-barrier method, contraceptive patch, male partner sterilization) before entry and throughout the study
* Body mass index (BMI) between 18 and 30 kilogram per square meter (kg/m^2) (inclusive), and body weight not less than 50 kilogram (kg)
* Systolic blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeter of mercury (mmHg) (inclusive) and diastolic blood pressure not more than 90 mmHg
* Comfortable with self-administration of intranasal medication and able to follow instructions provided
* A 12-lead electrocardiogram (ECG) consistent with normal cardiac conduction and function
* For Cohort 2, participants should have a history of allergic rhinitis and a positive prick test for grass pollen at screening
* For Cohort 2, participants must have a Total Nasal Symptoms Score (TNSS) greater than or equal to (>=) 6 with a nasal congestion score of >=2 (minimum for "moderate rhinitis") on at least one occasion while participants are in the ECC during screening

Exclusion Criteria:

* Current significant psychiatric (mental disorders) disorder including but not limited to psychotic (a person exhibiting mental illness), bipolar, major depressive or anxiety disorder
* Clinically significant medical illness including (but not limited to) cardiac arrhythmias (irregular heart beat) or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias [disorder of blood]), lipid abnormalities, significant pulmonary (having to do with the lungs) disease, including bronchospastic respiratory disease, diabetes mellitus (disorder in which there is decreased insulin in the body or the body's insulin is not effective, resulting in high blood sugar, increased thirst and urine, and many other side effects), renal or hepatic insufficiency, thyroid disease, neurologic disease, infection, hypertension or vascular disorders, kidney or urinary tract disturbances, sleep apnea (breathing problems while sleeping), myasthenia gravis (disorder that causes muscles to get tired quickly), or any other illness that the Investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Use of any prescription or nonprescription medication, within 14 days before the first scheduled dose of the study drug
* Anatomical or medical conditions that may delay delivery or absorption of study medication (for example. undergone facial reconstructions, structural or functional abnormalities of the nose or upper airway; obstructions or mucosal lesions [any visible local abnormality of the tissues of the skin] of the nostrils or nasal passages; undergone sinus [a depression or cavity formed by a bending or curving] surgery in the previous 2 years; or signs and symptoms of upper respiratory infection, rhinitis [Cohort 1 only], active allergies [Cohort 1 only], or has a history of frequent sinus infections or complications)
* Has an abnormal or deviated nasal septum (when the inner wall separating the two sides of the nose is off to one side) with any 1 or more of the following symptoms: blockage of 1 or both nostrils, nasal congestion (especially 1- sided), frequent nosebleeds, frequent sinus infections, noisy breathing during sleep, facial pain, headaches, and postnasal drip

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2014-06; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 0 (pre-dose), 7, 12, 22, 32, 40, 50 minutes; 1, 1.25, 1.5, 2, 3, 4, 6, 9, 12, 18, 24 and 30 hours after study drug administration
  The Cmax is the maximum plasma concentration.
Time to Reach Maximum Concentration (tmax) | 0 (pre-dose), 7, 12, 22, 32, 40, 50 minutes; 1, 1.25, 1.5, 2, 3, 4, 6, 9, 12, 18, 24 and 30 hours after study drug administration
  The tmax is time to reach the maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | 0 (pre-dose), 7, 12, 22, 32, 40, 50 minutes; 1, 1.25, 1.5, 2, 3, 4, 6, 9, 12, 18, 24 and 30 hours after study drug administration
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(0-last)/lambda(z), wherein AUC(0-last) is area under the plasma concentration time curve from time zero to last quantifiable time; C(0-last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Elimination Half-Life (t [1/2] Lambda) | 0 (pre-dose), 7, 12, 22, 32, 40, 50 minutes; 1, 1.25, 1.5, 2, 3, 4, 6, 9, 12, 18, 24 and 30 hours after study drug administration
  Elimination half-life (t [1/2] Lambda) is associated with the terminal slope (lambda [z]) of the semi logarithmic drug concentration-time curve, calculated as 0.693/lambda(z).
Number of participants with adverse events (AEs) and serious adverse events (SAEs) | Screening Up to 10 days after last study drug administration in Cohort 1 and Cohort 2
  An AE is any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non investigational) product and does not necessarily have a causal relationship with the treatment. An SAE is any untoward medical occurrence that meets any of the following conditions: results in death, is life threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, or is a congenital anomaly/birth defect.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Hanover, Germany

REFERENCES:
- [Derived] Zannikos P, Solanki B, De Meulder M, Badorrek P, Hohlfeld JM, Singh J. Pharmacokinetics of Nasal Esketamine in Patients with Allergic Rhinitis with and Without Nasal Decongestant Pretreatment and in Healthy Subjects with and Without Nasal Corticosteroid Pretreatment. Clin Pharmacokinet. 2023 Sep;62(9):1315-1328. doi: 10.1007/s40262-023-01273-z. Epub 2023 Jul 4. PMID 37402024